CLINICAL TRIAL: NCT01002989
Title: Assessment of the Oscillometric Measurement of the Ankle-brachial Index (ABI) With WatchBP Office ABI Device.
Brief Title: Validation of WatchBP Office Ankle-brachial Index (ABI) Function
Acronym: ABI
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Collaborators: Microlife (Industry)
Responsible Party: Principal Investigator, George S. Stergiou, Associate Professor of Medicine and Hypertension, University of Athens
Other Study IDs: Microlife ABI
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Hypertension
Keywords: ankle brachial index; WatchBP Office; oscillometric measurement
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All eligible patients: Subjects assessed for hypertension, were subjected to the measurement of ankle brachial index (ABI) by two methods:
  1. Doppler
  2. WatchBP Office oscillometric The order for performing the two methods was randomized.
  Interventions: Device: Doppler Ankle-Brachial Index measurement; Device: WatchBP Office Ankle-Brachial Index measurement.

INTERVENTIONS:
Device: Doppler Ankle-Brachial Index measurement — Measurement of the Ankle-Brachial Index by Doppler.
Device: WatchBP Office Ankle-Brachial Index measurement. — Measurement of Ankle-Brachial Index by WatchBP Office device.

SUMMARY:
Measurement of the ankle-brachial index (ABI) with the oscillometric device WatchBP Office will be assessed compared to the reference method (Doppler).

Ninety three adult subjects assessed for hypertension, treated or untreated, with complete study data were included. Data on the presence of cardiovascular (CV) disease and classical CV risk factors were recorded.

All the ABI measurements of each individual participant will be performed by the same observer in a randomized order (concerning Doppler and WatchBP)

DETAILED DESCRIPTION:
All study measurements were performed under standardized conditions in a quiet examination room with 10 min rest in the supine position before measurements. Ankle-brachial index (ABI) was measured manually by Doppler and automatically by the oscillometric device in randomized order by a single investigator. Manual Doppler ABI was measured according to the American Heart Association guidelines using a continuous wave Doppler device (Hadeco Bidop ES-100V3, Kawasaki, Japan) with a 8 MHz probe. Systolic blood pressure was defined with a standard mercury sphygmomanometer by the first Doppler flow signal while deflating the cuff from a suprasystolic level in brachial, dorsalis pedis and posterior tibial arteries. Systolic pressure was determined sequentially for brachial, dorsalis pedis and posterior tibial arteries for each side and ABI was calculated for each leg by dividing the highest ankle pressure to the highest arm pressure. Automated ABI measurement was performed using a validated oscillometric blood pressure monitor designed for professional use in the office (WatchBP Office device; Microlife, Widnau, Switzerland). This device allows automated simultaneous both arms or arm and leg blood pressure measurements and thereby the calculation of ABI. The ABI results are displayed on the device screen.

The study protocol included three steps: (i) an introductory familiarization automated ABI measurement, (ii) three simultaneous oscillometric both arms blood pressure measurements; in case of a consistent inter-arm difference ≥12 mmHg, the arm with the higher blood pressure was selected for the subsequent oscillometric ABI measurements (otherwise the right arm was used) and (iii) Doppler and automated ABI measurement in randomized order; Doppler ABI was measured once, whereas automated ABI calculation included triplicate simultaneous arm-leg measurements performed for each side. The occurrence of five sequential oscillometric errors was defined as a failure of the oscillometric device to measure ABI.

ELIGIBILITY:
Inclusion Criteria:

* Treated or untreated subjects assessed for hypertension

Exclusion Criteria:

* Atrial fibrillation
* Incompressible ankle arteries

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects assessed for hypertension including those with other cardiovascular risk factors
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George S Stergiou, Assoc. Prof., Principal Investigator — Hypertension Center, University of Athens, Greece
Locations (1):
- Hypertension Center, Sotiria Hospital, Athens, Greece

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with various cardiovascular risk factors attending a hypertension or a diabetes outpatient clinic during the period 10/2009-06/2010 were invited to participate in the study
Groups:
- Hypertensives: Subjects assessed for hypertension underwent manual Doppler ABI measurement using a continuous wave Doppler device (Hadeco Bidop ES-100V3, Kawasaki, Japan) with a 8 MHz probe and automated ABI measurement using a validated oscillometric blood pressure monitor designed for professional use in the office (WatchBP Office device; Microlife, Widnau, Switzerland).
Period: Overall Study
Arm/Group | Hypertensives
Started | 98
Completed | 93
Not Completed | 5
Not completed — exclusion criteria, no consent | 5

BASELINE CHARACTERISTICS:
Arm/Group | Hypertensives
Number analyzed (Participants) | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 44
Age Continuous [Mean (Standard Deviation); unit: years] | 62.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 61
Region of Enrollment [Number; unit: participants]
  Greece | 98
Mean Doppler ABI [Mean (Standard Deviation); unit: ratio] | 1.08 (0.17)
Watch BP Office minus Doppler Ankle-Brachial Index (ABI) difference [Mean (Standard Deviation); unit: ratio] | 0.03 (0.11)
Mean Watch BP Office ABI [Mean (Standard Deviation); unit: ratio] | 1.11 (0.17)

OUTCOME MEASURES:

1. Primary Outcome: Watch BP Office Minus Doppler Ankle-Brachial Index Difference
Description: The validation process consisted of two parts: (i) measurement validation, which compared Doppler and Watch BP Office ABI values and assessed their association, and (ii) clinical validation, which compared the diagnosis of peripheral artery disease (PAD) by the two methods and assessed the association of Watch BP Office and Doppler ABI values with cardiovascular risk factors.
Time Frame: once (cross-sectional)
Population: Patients with various cardiovascular risk factors attending a hypertension or a diabetes outpatient clinic were invited to participate in the study. Subjects with atrial fibrillation or incompressible ankle arteries (ABI ≥1.4) were excluded.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Hypertensives
Number analyzed (Participants) | 93
ratio | 0.03 (0.11)

2. Secondary Outcome: Agreement Between the Two Methods in Peripheral Artery Disease (PAD) Diagnosis
Description: This outcome measure represents what percentage of the patients diagnosed with PAD using Doppler ABI method (reference method) were diagnosed with PAD using WatchBP Office ABI method. It also represents in what percentage of the patients in whom PAD was excluded with Doppler ABI method (reference method), PAD was excluded using WatchBP Office ABI method as well.
Time Frame: Once (cross-sectional)
Measure: Number; unit: Percentage of participants
Arm/Group | Hypertensives
Number analyzed (Participants) | 93
Percentage of participants | 95

3. Primary Outcome: Mean Doppler Ankle-Brachial Index
Time Frame: once (cross-sectional)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Hypertensives
Number analyzed (Participants) | 93
ratio | 1.08 (0.17)

4. Primary Outcome: Mean Watch BP Office Ankle-Brachial Index
Time Frame: once (cross-sectional)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Hypertensives
Number analyzed (Participants) | 93
ratio | 1.11 (0.17)

ADVERSE EVENTS:
Arm/Group | Hypertensives
Serious Adverse Events (participants affected / at risk) | 0/93
Other Adverse Events (participants affected / at risk) | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No